CLINICAL TRIAL: NCT04693351
Title: A Randomized, Double-Blind, Placebo- Controlled Trial of Adjunctive Troriluzole in Obsessive Compulsive Disorder
Brief Title: Efficacy and Safety Study of Adjunctive Troriluzule in Obsessive Compulsive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV4157-303
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder (OCD)
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Troriluzole (Experimental): Troriluzole- 2 100mg capsules once daily for the first two weeks. Troriluzole- 2 140mg capsules once daily from week two through week ten.
  Interventions: Drug: Troriluzole
- Placebo (Placebo Comparator): Placebo- 2 100mg capsules once daily for the first two weeks. Placebo- 2 140mg capsules once daily from week two through week ten.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Troriluzole — Two 100mg capsules daily for first two weeks and then two 140mg capsules daily from week 2 through week ten.
  Arms: Troriluzole
Drug: Placebo — Two 100mg capsules daily for first two weeks and then two 140mg capsules daily from week 2 through week ten.
  Arms: Placebo

SUMMARY:
The study's purpose its to evaluate the efficacy and safety of troriluzole as adjunctive therapy compared to placebo in subjects with Obsessive Compulsive Disorder (OCD)

ELIGIBILITY:
Key Inclusion Criteria:

1. Primary diagnosis of obsessive-compulsive disorder (OCD) as per Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition as confirmed by the MINI at screening; the duration of the subjects illness must be ≥ 1year
2. An inadequate response to current Standard of Care medication defined as selective serotonin reuptake inhibitor (excluding fluvoxamine) or clomipramine treatment at an adequate and stable dose for at least 8 weeks prior to screening and at least 12 weeks at baseline (adequate dose defined by USPI labeling); an inadequate response too current standard of car base on the YBOCS score.
3. Determined by the investigator to be medically stable at baseline/ randomization as assessed by medical history, physical examination, laboratory test results, and electrocardiogram testing. Subjects must be physically able and expected to complete the trail as designed.

Key Exclusion Criteria:

1. Subjects with a history of more than two (2) previous failed or inadequate treatment classes given for an adequate duration at an adequate dose as defined by the MGH-TRQ-OCD.
2. Current or prior history of: bipolar I or II disorder, schizophrenia or other psychotic disorders, schizoaffective disorder, autism or autism spectrum disorders, borderline personality disorder, antisocial personality disorder, Tourette's disorder, body dysmorphic disorder, hoarding disorder, or psychosurgery, Deep Brain Stimulation (DBS) or Electroconvulsive Therapy (ECT); or general medical condition that may confound safety and/or efficacy results.
3. Previous treatment in a study with troriluzole

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
The total score on the Yale-Brown Obsessive Compulsive Disorder (YBOCS) | Change in total score from baseline, assessed at screening, baseline, week 4, 8 &10
  Improvement is measured by a lower total score

SECONDARY OUTCOMES:
Frequency of SAEs and AEs leading discontinuation | From Screening through Study completion, up to 10 weeks
  Percent difference between troriluzole vs placebo treatment emergent adverse events
Improvement in function disability as assessed by the change in the Sheehan Disability Scale (SDS) | From baseline through study completion (up to 10 weeks)
  Change is measured as "mild" or "moderate" on the SDS
Improvement in global functioning responses as assessed on the CGI-I scale. | From baseline through study completion (up to 10 weeks)
  Change is measured as "much improved" or very much improved" on the CGI-I scale.

CONTACTS AND LOCATIONS:
Locations (89):
- United States (49):
  - Alea Research, Phoenix, Arizona
  - ProScience Research Group, Culver City, California
  - Kaizen Brain Center, La Jolla, California
  - Om Research LLC, Lancaster, California
  - CalNeuro Research Group, Los Angeles, California
  - Lumos Clinical Research Center, LLC, San Jose, California
  - Velocity Clinical Research, Santa Ana, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Mountain View Clinical Research, Denver, Colorado
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Topaz Clinical Research, Apopka, Florida
  - CNS Research of Coral Springs, Coral Springs, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - University of Florida Department of Psychiatry, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Med-Care Research, Miami, Florida
  - Ezy Medical Research, Co., Miami, Florida
  - Advanced Research for Health Improvement, Naples, Florida
  - Harmony Clinical Research, North Miami Beach, Florida
  - dTMS Center LLC, Palm Beach, Florida
  - DMI Research, Pinellas Park, Florida
  - CenExel iResearch, Decatur, Georgia
  - Renew Health Clinical Research, LLC, Snellville, Georgia
  - University of Chicago Department of Psychiatry & Behavioral Neuroscience, Chicago, Illinois
  - AMR-Baber Research, Inc., Naperville, Illinois
  - Collective Medical Research, Overland Park, Kansas
  - Continental Clinical Solutions, LLC, Towson, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - Boeson Research, Missoula, Montana
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Manhattan Behavioral Medicine, PLLC, New York, New York
  - Richard H. Weisler, MD PA & Associates, Raleigh, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - American Clinical Research Institute (ACRI), Dayton, Ohio
  - American Research Institute (ACRI), Kettering, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Donald J. Garcia Jr., MD PA, Austin, Texas
  - Inquest Clinical Research, Baytown, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Clinical Trial Network, Houston, Texas
  - AIM Trials, Plano, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Woodstock Research Center, Woodstock, Vermont
- Canada (7):
  - University of Calgary, Calgary, Alberta
  - Chatham-Kent Clinical Trials Research Centre, Chatham, Ontario
  - McMaster University, Hamilton Health Sciences, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - START Clinic for Mood and Anxiety Disorders, Toronto, Ontario
  - University of Toronto / Centre for Addiction and Mental Health (CAMH), Toronto, Ontario
- China (11):
  - Beijing HuiLongGuan Hospital, Beijing, Changping District
  - Peking University Sixth Hospital, Beijing, Haidian District
  - Hangzhou Seventh People's Hospital, Hangzhou, Hangzhou City
  - Tianjin Anding Hospital, Tianjin, Hexi District
  - The Second Xiangya Hospital of Central South University, Xiangya, Hunan
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - Shanghai Mental Health Center, Shanghai, Minhang District
  - Wuhan Mental Health Center, Wuhan, Qiaokou District
  - The First Affiliated Hospital of Jinan University, Guangzhou, Tianhe District
  - Mental Health Center, West China Hospital, Sichuan University, Chengdu, Wuhou District
  - First Hospital of Hebei Medical University, Shijiazhuang, Yuhua District
- Italy (4):
  - ASST FBF SACCO - Ospedale Universitario Luigi Sacco, Milan
  - University School of Medicine of Napoli Federico II, Naples
  - University of Pisa, Pisa
  - University of Turin - university hospital san luigi gonzaga, Turin
- Netherlands (2):
  - Amsterdam UMC, locatie AMC, Amsterdam
  - Leiden University Medical Center (LUMC), Leiden
- Spain (6):
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Centro de Salud Mental La Corredoria, Oviedo
  - Centro de Salud San Juan, Salamanca
  - Hospital Álvaro Cunqueiro, Vigo
- United Kingdom (10):
  - MAC Clinical Research, Stockton-on-Tees, County Durham
  - Stemax Consult - Healthcare Services Ltd, Stony Stratford, Northamptonshire
  - MAC Clinical Research - South Staffordshire, Cannock, South Staffordshire
  - MAC Clinical Research-Lancashire, Blackpool
  - MAC Clinical Research, Leeds
  - MAC Clinical Research -- Merseyside, Liverpool
  - Greater Manchester Mental Health NHS Foundation Trust, Manchester
  - Bioluminux Ltd, Milton Keynes
  - Kingshill Research Centre, Swindon
  - MAC Clinical Research-- South Yorkshire, Tankersley